CLINICAL TRIAL: NCT00022464
Title: A Phase II Study Of CCI-779 (NSC 683864) In Metastatic Melanoma
Brief Title: CCI-779 in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068820; U01CA063265 (NIH); P30CA033572 (NIH); CHNMC-PHII-27; CHNMC-IRB-99167; NCI-29
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — temsirolimus

INTERVENTIONS:
Drug: temsirolimus

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of CCI-779 in treating patients who have metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the anti-tumor activity of CCI-779, in terms of progression-free survival, in patients with metastatic melanoma.
* Determine the toxic effects of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive CCI-779 IV over 30 minutes on day 1. Courses repeat every 7 days in the absence of disease progression or unacceptable toxicity.

Patients are followed for survival.

PROJECTED ACCRUAL: Approximately 40-50 patients will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic melanoma that is incurable by surgery, radiotherapy, or limb perfusion
* Measurable disease

  * At least 20 mm by conventional techniques OR
  * At least 10 mm by spiral CT scan
  * The following are not considered measurable:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
    * Abdominal masses not confirmed and followed by imaging techniques
    * Cystic lesions
* Progressive disease
* No prior or concurrent CNS metastasis

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* More than 4 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin normal
* AST and ALT no greater than 2.5 times upper limit of normal
* Cholesterol no greater than 350 mg/dL (lipid-lowering therapy allowed)
* Triglycerides no greater than 300 mg/dL except for hydroxymethyl-glutaryl-coenzyme A reductase inhibitors

Renal:

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No prior allergic reactions to compounds of similar chemical or biological composition to study drug
* No ongoing or active infection
* No seizure disorder
* No autoimmune disease
* No psychiatric illness or social situation that would preclude study
* No other concurrent uncontrolled illness that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No more than 1 prior adjuvant biological therapy regimen
* No more than 1 prior biological therapy regimen for advanced disease
* At least 6 months since prior biological therapy or biochemotherapy and recovered
* Prior isolated limb perfusion with biological agent allowed if not to sole site of disease

Chemotherapy:

* See Biologic therapy
* Prior isolated limb perfusion with chemotherapy allowed if not to sole site of disease
* No more than 1 prior chemotherapy-containing regimen for advanced disease, regardless of adjuvant therapy

  * May be in addition to 1 prior biologic regimen for advanced disease OR
  * May have had 1 prior biochemotherapy regimen for advanced disease
* At least 3 weeks since prior chemotherapy and recovered

Endocrine therapy:

* At least 1 week since prior dexamethasone
* No concurrent glucocorticosteroid therapy

Radiotherapy:

* See Disease Characteristics

Surgery:

* See Disease Characteristics

Other:

* At least 1 week since prior phenobarbital, phenytoin, carbamazepine, or rifampin
* At least 3 weeks since other prior agents to treat malignancy
* At least 3 weeks since prior investigational agents
* No other concurrent investigational agents
* No concurrent drugs that are metabolized by or alter the level of cytochrome P450-3A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-06; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim A. Margolin, MD, Study Chair — City of Hope Comprehensive Cancer Center
Locations (21):
- United States (18):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - City of Hope Medical Group, Pasadena, California
  - University of California Davis Cancer Center, Sacramento, California
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Evanston Northwestern Health Care - Evanston Hospital, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - LaGrange Memorial Hospital, LaGrange, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - North Shore University Hospital, Manhasset, New York
  - Weill Medical College of Cornell University, New York, New York
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
- Canada (3):
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Result] Margolin K, Longmate J, Baratta T, Synold T, Christensen S, Weber J, Gajewski T, Quirt I, Doroshow JH. CCI-779 in metastatic melanoma: a phase II trial of the California Cancer Consortium. Cancer. 2005 Sep 1;104(5):1045-8. doi: 10.1002/cncr.21265. PMID 16007689